CLINICAL TRIAL: NCT03036566
Title: Clinical Evaluation of Chairside Computer Assisted Design/Computer Assisted Machining (CAD/CAM) Lithium Disilicate Fixed Partial Dentures (FPD)
Brief Title: Lithium Disilicate (CAD/CAM) Fixed Partial Dentures (FPD) Clinical Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Loss of funding due to COVID-19
Sponsor: University of Michigan (Other)
Collaborators: Ivoclar Vivadent AG (Industry)
Responsible Party: Principal Investigator, Dennis J. Fasbinder, DDS, Clinical Professor, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HUM00081086
Record Dates: First submitted 2017-01-26; First posted 2017-01-30 (Estimated); Results first posted 2023-04-05 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Missing Tooth
MeSH Terms: conditions — Anodontia | interventions — Denture, Partial, Fixed

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Bridge (Experimental): Three unit high strength ceramic (lithium disilicate/emaxCAD by Ivoclar) bridges replacing a single tooth.
  Interventions: Device: Lithium disilicate ceramic (Ivoclar)

INTERVENTIONS:
Device: Lithium disilicate ceramic (Ivoclar) — Three unit high strength ceramic bridges replacing a single tooth.
  Other Names: fixed partial denture

SUMMARY:
This investigation will be a clinical trial to study the performance of a high strength ceramic material for bridges to replace missing teeth. The ceramic material has been approved by the FDA for patient treatment. A computer technique will be used to make the bridges. The bridges will be cemented using an adhesive resin cement (MultiLink Automix/Ivoclar). The bridges are planned be evaluated for clinical performance at 6 months, 1 year, 2 years, 3 years, and if funding permits, 4 years, and 5 years. The purpose of the study is to measure how well the high strength bridges function over an extended period of time.

DETAILED DESCRIPTION:
The study will be composed of 30 bridges placed in adult patients that have been identified as requiring replacement of a single tooth. All the bridges will be made from the same high strength ceramic material (emaxCAD/Ivoclar) using a computer to make the entire bridge. All the crowns will be cemented using the most current marketed version of the manufacturer's adhesive resin cement (MultiLink Automix/Ivoclar). At each recall appointment an evaluation of the bridge will be completed as well as clinical photographs, an intraoral digital scan, and impression of the bridge. The purpose of the study is to measure how well the high strength bridges function over an extended period of time.

ELIGIBILITY:
Inclusion Criteria:

* missing one anterior or premolar tooth that is appropriate for replacement with a bridge. The second premolar tooth will be the most distal tooth acceptable as a pontic for inclusion in the study.
* healthy periodontal status for the adjacent abutment teeth with 1:1 crown:root ratio
* abutment teeth must be asymptomatic prior to treatment
* Endodontically treated teeth will be acceptable for abutments as long as nonmetallic cores can be placed to retain the FPD since the lithium disilicate will be bonded to the abutments.
* no more than one bridge will be placed per patient. If a patient presents with more than one missing teeth acceptable for the study, premolar teeth will be included prior to anterior teeth. Each bridge will be three units and include only one missing tooth.

Exclusion Criteria:

* sensitive abutment teeth
* teeth with a history of direct or indirect pulp capping procedures
* patients with significant untreated dental disease to include periodontitis and caries
* pregnant or lactating women
* patients with allergies to any material in the study
* patients unable to return for recall appointments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-03; Primary Completion 2020-03-05 (Actual); Study Completion 2020-03-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dennis J Fasbinder, DDS, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Bridge
Started | 30
Completed | 27
Not Completed | 3
Not completed — Lost to Follow-up | 3

BASELINE CHARACTERISTICS:
Arm/Group | Bridge
Number analyzed (Participants) | 30
Age, Customized [Count of Participants; unit: Participants] — Age was not collected from any participant.
  Participants | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 11
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Bridge Failure
Description: Bridge failure includes fracture of the bridge or loss of the bridge requiring placement of a new bridge at any time between delivery and five years.
Time Frame: from delivery of the bridge up to 5 years
Measure: Number; unit: number of bridges
Arm/Group | Bridge
Number analyzed (Participants) | 30
number of bridges | 2

2. Secondary Outcome: Bridge Loss of Retention
Description: Loss of retention is measured as detachment of the bridge from the teeth without fracture of the bridge requiring recementation of the bridge.
Time Frame: from delivery of the bridge up to 5 years
Measure: Number; unit: number of bridges
Arm/Group | Bridge
Number analyzed (Participants) | 30
number of bridges | 0

3. Secondary Outcome: Number of Bridges Associate With Tooth Sensitivity
Description: Tooth Sensitivity is evaluated as either "0" if the subject reports that there is NO sensitivity for either tooth with the study bridge, or "1" if the subject reports that there IS tooth sensitivity to hot/cold or biting pressure for either tooth supporting the bridge. The better outcome is to have NO tooth sensitivity.
Time Frame: from delivery of the bridge up to 5 years
Population: number of bridges
Measure: Number; unit: number of bridges
Arm/Group | Bridge
Number analyzed (Participants) | 30
number of bridges | 0

4. Secondary Outcome: Number of Bridges Associated With Margin Staining
Description: Margin Staining is evaluated as either "0" if there is NO staining at the crown margin where it meets the tooth for either tooth supporting the bridge, or "1" if there IS staining at the crown margin where it meets the tooth for either tooth supporting the bridge. The better outcome is to have NO margin staining.
Time Frame: from delivery of the bridge up to 5 years
Population: number of bridges
Measure: Number; unit: number of bridges
Arm/Group | Bridge
Number analyzed (Participants) | 30
number of bridges | 3

ADVERSE EVENTS:
Time Frame: 5 years
Arm/Group | Bridge
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-05-23): https://cdn.clinicaltrials.gov/large-docs/66/NCT03036566/Prot_SAP_000.pdf